CLINICAL TRIAL: NCT02289170
Title: A Randomized, Double-blind, Multicenter, Parallel Designed Clinical Study to Evaluate the Safety and Efficacy of Heating and Cooling Combination Therapeutic Device(OCH-S100) in Patients With Chronic Low Back Pain
Brief Title: Clinical Study to Evaluate the Safety and Efficacy of Heating and Cooling Combination Therapeutic Device(OCH-S100)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eun Jung Kim (Other)
Collaborators: Ministry of Health & Welfare, Korea (Other Government)
Responsible Party: Sponsor-Investigator, Eun Jung Kim, Clinical trial Chief of Research, DongGuk University
Organization: DongGuk University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OCH-S100-2014; HI11C2135 (Other Grant/Funding Number: The Korea Health Industry Development Institute)
Record Dates: First submitted 2014-10-14; First posted 2014-11-13 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Chronic Low Back Pain
Keywords: Chronic low back pain; Heating and cooling combination therapeutic device; Heating and cooling combination therapy; Contrast therapy
MeSH Terms: interventions — Cryotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Heating and cooling combination therapy (Experimental): The patients in this group received heating and cooling combination therapy by a certified Korean Medicine Doctor with more than 6 years of oriental medicine college education and 2 years of clinical experience. Doctor press 8 acupuncture points which is treated in LBP patients and select the most painful 2 acupuncture points. Device's probe is attached to the acupuncture points in 15 minutes. Probe's temperature is changed 5 cycles from maximum 45℃ to minimum 15℃.
  Interventions: Device: Heating and cooling combination therapy
- Sham heating and cooling therapy (Sham Comparator): The patients in this group received sham heating and cooling combination therapy in same conditions of treatment group except the temperature. Before the treatment begin, caregiver measure the patient's skin temperature. Then probe's temperature is changed 5 cycles from 1℃ over the skin temperature to 1℃ under the skin temperature.
  Interventions: Device: Sham heating and cooling therapy

INTERVENTIONS:
Device: Heating and cooling combination therapy — The treatment was applied 10 times for 4 weeks. Most painful 2 points in 8 acupuncture points(both side of Bladder meridian23 (BL23), BL24, BL25, BL26) were used for all the patients assigned to this group.
  Other Names: OCH-S100
  Arms: Heating and cooling combination therapy
Device: Sham heating and cooling therapy — The treatment was applied 10 times for 4 weeks. The sham heating and cooling combination therapy was applied on the 2 of 8 same acupuncture points as in the treatment group.
  Other Names: OCH-S100
  Arms: Sham heating and cooling therapy

SUMMARY:
The purpose of this study is to verify the efficacy and safety of heating and cooling combination therapeutic device (OCH-S100) for patients with chronic low back pain (LBP).

DETAILED DESCRIPTION:
The investigators targeted the patients with chronic LBP. After treatment in 2 groups - real heating and cooling combination treatment and sham heating and cooling combination treatment - the investigators will compare the effects of pain relief and improvement in disability and range of motion of lumbar region. So the investigators will confirm the efficacy of heating and cooling combination therapy, and further the best treatment method. In addition, the investigators are going to evaluate the safety of abnormal reaction during the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. At least 20 years of age, but below 75 years of age
2. Low back pain in the last 3 months or more
3. Low back pain rated over 40 mm on a 100 mm Visual Analog Scale (VAS)
4. Those who are reliable and willing to cooperate in this test, and obey the restrictions for the treatment period.
5. An understanding of the objectives, methods and efficacy of the clinical trial, and willingness in completing the consent form.

Exclusion Criteria:

1. Trauma to or surgery on the lumbar region within 6 months prior to enrollment
2. Low back pain accompanied by sciatica
3. Systematic disease, and severe dysfunction due to the medical illness (e.g. cancer, infection, etc.)
4. A history of medication, oriental medical treatment, physiotherapy for treating low back pain within the last 4 weeks
5. Neurological disease, such as topical or whole body hypoesthesia in temperature sensation (e.g. stroke, peripheral neuropathy, etc.)
6. Hypersensitivity in heating and cooling stimulation
7. Pregnant and lactating women
8. Participate in the other clinical trials within the last 3 months or after enroll this trial
9. When researchers evaluate that it is not appropriate to participate in this clinical test

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in 100mm Pain Visual Analogue Scale (VAS) | at baseline and 4 4 weeks later from baseline
  The patient is asked to indicate their perceived pain intensity along a 100 mm horizontal line, where '0' represents 'no pain' and '100', 'unbearable pain'

SECONDARY OUTCOMES:
Change from baseline in 100mm Pain Visual Analogue Scale (VAS) | estimately every 2.8 days from baseline to 4 weeks later, and 4 weeks later from the end of treatment
  The patient is asked to indicate their perceived pain intensity along a 100 mm horizontal line, where '0' represents 'no pain' and '100', 'unbearable pain'
Change from baseline in Korean Oswestry disability index (KODI) | at baseline, 2 weeks and 4 weeks later from baseline, and 4 weeks later from the end of treatment
  KODI is checked by the patients. KODI is a questionnaire to measure the back-related disability. KODI consists of combination of physical and social restriction through 9 questions covering different dimensions of daily living.
Change from baseline in Korean Roland Morris Disability Questionnaire (KRMDQ) | at baseline, 2 weeks and 4 weeks later from baseline, and 4 weeks later from the end of treatment
  KRMDQ is checked by the patients. KRMDQ is a questionnaire to measure the back-related disability. KRMDQ consists of 24 questions answered yes or no.
Change from baseline in Traditional Medicine Back pain Questionnaire (TMBQ) | at baseline, 2 weeks and 4 weeks later from baseline, and 4 weeks later from the end of treatment
  TMBQ is checked by the patients. TMBQ is a questionnaire to measure the back-related disability in aspect of oriental medicine.
Change from baseline in Modified schöber test | at baseline, 2 weeks and 4 weeks later from baseline, and 4 weeks later from the end of treatment
  Modified schöber test measures the flexion range of motion of lumbar spine. First, investigator marks the point at patients' lumbosacral junction. Then also marks the points at upper 10cm and lower 5cm of the former point in standing position. After marking the 3 points, patients bend anteriorly as best he or she can. Then, investigator measures the length of the latter 2 points.
Change from baseline in Finger-to-floor distance | at baseline, 2 weeks and 4 weeks later from baseline, and 4 weeks later from the end of treatment
  Finger-to-floor distance measures the flexion range of motion of lumbar spine. Patients stand on the box which height is 20cm. Then, patients bend anteriorly in extension of knee and upper limb. Investigator measures the length from floor to 3rd finger.
Change from baseline in Finger-to-thigh distraction | at baseline, 2 weeks and 4 weeks later from baseline, and 4 weeks later from the end of treatment
  Finger-to-thigh distraction measures the lateral bending range of motion of lumbar spine. Patients stand on the box which height is 20cm. Then, patients bend laterally in extension of knee and upper limb. Investigator measures the length from floor to 3rd finger.
Adverse Events | estimately every 2.8 days from baseline to 4 weeks later, and 4 weeks later from the end of treatment
  Any unpredicted symptoms were checked at each follow up visit and if any, the symptom, time of occurrence, and length of duration were recorded and reported.

CONTACTS AND LOCATIONS:
Overall Officials: Seung Deok Lee, Ph.D., Principal Investigator — Donnguk University Oriental Medical center
Locations (1):
- Donnguk University Oriental Medical Hospital, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Kim EJ, Choi YD, Lim CY, Kim KH, Lee SD. Effect of heating and cooling combination therapy on patients with chronic low back pain: study protocol for a randomized controlled trial. Trials. 2015 Jun 26;16:285. doi: 10.1186/s13063-015-0800-4. PMID 26112148